CLINICAL TRIAL: NCT01287507
Title: Oral Lactoferrin Prophylaxis to Prevent Sepsis and Necrotising Enterocolitis of Very Low Birth Weight Neonates in Neonatal Intensive Care Unit and Effect on T-regulatory Cells.
Brief Title: Lactoferrin Prophylaxis in VLBW and Regulator T-cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ilke Mungan Akin, Neonatologist, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lactoferrin
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Late Onset Neonatal Sepsis; Necrotising Enterocolitis; Very Low Birth Weight Infants
Keywords: VLBW, NEC, Late onset sepsis
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing | interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In born VLBW infants with parental consent form signed will be given oral saline daily as placebo until discharge
  Interventions: Dietary Supplement: Lactoferrin (bovine origin)
- Lactoferrin (Experimental): In born VLBW infants with parental consent form signed will be given oral bovine lactoferrin daily until discharge
  Interventions: Dietary Supplement: Lactoferrin (bovine origin)

INTERVENTIONS:
Dietary Supplement: Lactoferrin (bovine origin) — Bovine lactoferrin 200 mg/daily, given with either human milk or preterm formula

SUMMARY:
The aim of the study is to evaluate whether oral administration of 200 mg/day lactoferrin (LF) to very low birth weight infants reduces late onset sepsis and necrotising enterocolitis and the effect of LF on regulatory T cells.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants
* Gestational age < 32 weeks
* Birth weight < 1500 g
* Parental consent

Exclusion Criteria:

* Congenital abnormalities
* Severe perinatal asphyxia

Ages: 15 Minutes to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
late onset sepsis | from birth to discharge from NICU
  The effect of oral Lactoferrin prophylaxis on the number of culture proven sepsis attacks in very low birth weight infants during their hospitalization in neonatal intensive care unit. Sterile blood, urine and cerebrospinal fluid samples will be obtained in case of clinical symptoms of sepsis for culture.
Necrotising enterocolitis | from birth to discharge from NICU
  The effect of oral Lactoferrin prophylaxis on severe necrotising enterocolitis (NEC) (Bell's stage 2 and 3) in very low birth infants during the hospitalization period in Neonatal intensive care unit. In case of feeding intolerance, abdominal distention and findings of ileus with clinical deterioration, patient will be evaluated for thrombocytopenia, metabolic acidosis, hyponatremia, blood in stool and radiological findings of NEC. Staging will be performed with clinical, laboratory and radiological findings.
Effect on T regulatory cells | at discharge
  FOXP3 expression on CD4+CD25+ T cells

SECONDARY OUTCOMES:
Safety of lactoferrin in VLBW infants | during the oral use of lactoferrin
  the effect oral lactoferrin use on feeding tolerance, abdominal distension, vomiting and gastric residuals
duration of hospitalization | from birth to discharge from neonatal intensive care unit
  the effect of oral lactoferrin on the duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Arsan, Prof, Study Chair — Anlara University Chief of Neonatology
Locations (1):
- Ankara University School of Medicine Department of Pediatrics, NICU, Ankara, Turkey (Türkiye)